CLINICAL TRIAL: NCT06816030
Title: An Open-label Study to Characterize the Pharmacokinetics, Safety and Tolerability of Single and Multiple Oral Doses of MK-4482 in Chinese Healthy Male Participants
Brief Title: A Clinical Study of MK-4482 in Chinese Healthy Male Participants (MK-4482-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4482-009; MK-4482-009 (Other: MSD)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir

STUDY DESIGN:
Intervention Model Description: Sequential model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MK-4482 (Experimental): Participants in period 1 received, MK-4482 800 mg single oral dose in the morning on Day 1. Participants in period 2 received, MK-4482 800mg oral dose administered every 12 hours (Q12H) on Day 1 through Day 6 for11 doses.
  Interventions: Drug: MK-4482

INTERVENTIONS:
Drug: MK-4482 — Participants in period 1 received, MK-4482 800 mg single oral dose in the morning on Day 1. Participants in period 2 received, MK-4482 800mg oral dose administered every 12 hours (Q12H) on Day 1 through Day 6 for11 doses.

SUMMARY:
The goal of the study is to learn what happens to MK-4482 after single and multiple doses in healthy Chinese participants over time. Researchers also want to learn about the safety of MK-4482, including how well people tolerate it.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

- Has a Body Mass Index (BMI) of 19 to 24 weight (kg)/height (m)2, inclusive, and body weight of ≥ 50 kg at the screening visit.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a history of clinically significant abnormalities or diseases.
* Has history of cancer.
* Has a history of significant multiple and/or severe allergies.
* Had any major surgery.
* Has participated in another investigational study within 3 months prior to the screening visit.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male adult participants of Chinese descent
Enrollment: 16 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
The Maximum Observed Plasma Concentration (Cmax) After Single Oral Dose of MK-4482 in Period 1 | At designated time points up to 72 hours post-dose
  Cmax of N-hydroxycytidine (NHC) after a single oral dose of MK-4482 in period 1.
Time to Reach Maximum Observed Plasma Concentration (Tmax ) After Single Oral Dose of MK-4482 in Period 1. | At designated time points up to 72 hours post-dose
  Tmax of NHC following single oral dose of MK-4482 in period 1.
Elimination Half Life (T1/2) After Single Oral Dose of MK-4482 in Period 1 | At designated time points up to 72 hours post-dose
  T1/2 is defined as the time required for the concentration or amount of NHC in the body to be reduced by one-half after a single oral dose of MK-4482 in period 1.
Apparent Total Clearance (CL/F) After Single Oral Dose of MK-4482 in Period 1 | At designated time points up to 72 hours post-dose
  CL/F of NHC from plasma after single oral dose of MK-4482 in period 1.
Apparent Volume of Distribution (Vz/F) After Single Oral Dose of MK-4482 in Period 1 | At designated time points up to 72 hours post-dose
  Vz/F of NHC during terminal phase after single oral dose of MK-4482 in period 1.
Area Under the Plasma Concentration-time Curve From Time 0 to 12 Hours Post-dose (AUC0-12hr) After Single Oral Dose of MK-4482 in Period 1 | At designated time points up to 72 hours post-dose
  This is a measure of the average amount of NHC in the plasma over a period of 12 hours after single oral dose of MK-4482 in period 1.
Area Under the Plasma Concentration-time Curve From Time Zero to Last Measurable Concentration (AUC0-last) After Single Oral Dose of MK-4482 in Period 1 | At designated time points up to 72 hours post-dose
  AUC0-last of NHC following a single oral dose of MK-4482 in period 1.
Area Under The Plasma Concentration Versus Time Curve From Time Zero (pre-dose) to Extrapolated Infinite Time (AUC0-inf) After Single Oral Dose of MK-4482 in Period 1 | At designated time points up to 72 hours post-dose
  AUC0-inf of NHC after single oral dose of MK-4482 in period 1.
The Maximum Observed Plasma Concentration (Cmax) After Multiple Oral Doses of MK-4482 in Period 2 | At designated time points up to 72 hours post-dose
  Cmax of NHC after multiple oral doses of MK-4482 in period 2.
Time to Reach Maximum Observed Plasma Concentration (Tmax ) After Multiple Oral Doses of MK-4482 in Period 2 | At designated time points up to 72 hours post-dose
  Tmax of NHC following multiple oral doses of MK-4482 in period 2.
Elimination Half Life (T1/2) After Multiple Oral Doses of MK-4482 in Period 2 | At designated time points up to 72 hours post-dose
  T1/2 is defined as the time required for the concentration or amount of NHC in the body to be reduced by one-half after multiple oral doses of MK-4482 in period 2.
Clearance at Steady State (CLss/F) After Multiple Oral Doses of MK-4482 in Period 2 | At designated time points up to 72 hours post-dose
  CLss/F of plasma NHC following multiple doses of MK-4482 in period 2.
Apparent Volume of Distribution (Vz/F) After Multiple Oral Doses of MK-4482 in Period 2 | At designated time points up to 72 hours post-dose
  Vz/F of NHC during terminal phase after multiple doses of MK-4482 in period 2.
Area Under the Plasma Concentration-time Curve From Time 0 to 12 Hours Post-dose (AUC0-12hr) After Multiple Oral Doses of MK-4482 in Period 2 | At designated time points up to 72 hours post-dose
  This is a measure of the average amount of NHC in the plasma over a period of 12 hours after multiple oral doses of MK-4482 in period 2.
The Minimum Concentration (Ctrough) After Multiple Oral Doses of MK-4482 in Period 2 | At designated time points up to 72 hours post-dose
  Ctrough of NHC that occurred following multiple doses of MK-4482 in period 2.
Accumulation Ratio on Cmax After Multiple Oral Doses of MK-4482 in Period 2 | At designated time points up to 72 hours post-dose
  The maximum concentration at steady state following multiple doses of MK-4482 in period 2 divided by the maximum concentration following the initial dosing in Period 1.
Accumulation Ratio on AUC0-12hr After Multiple Oral Doses of MK-4482 | At designated time points up to 72 hours post-dose
  The AUC0-12hr at steady state following multiple doses of MK-4482 in period 2 divided by the AUC0-12hr following the initial dosing in Period 1.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to ~ 5.5 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to ~ 5.5 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Peking University Third Hospital (Site 0001), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com